CLINICAL TRIAL: NCT00599703
Title: Reorganization of Language Function in Patients With Brain Tumors
Brief Title: Language Function in Patients With Brain Tumors
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Andrei Holodny, M.D., Memorial Sloan-Kettering Cancer Center
Other Study IDs: 05-043
Record Dates: First submitted 2008-01-11; First posted 2008-01-24 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Brain Cancer; CNS Cancer
MeSH Terms: conditions — Brain Neoplasms; Central Nervous System Neoplasms | interventions — Lead

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: neurosurgical patients
  Interventions: Other: fMRI Scan, pre- and post language evaluation

INTERVENTIONS:
Other: fMRI Scan, pre- and post language evaluation — All subjects will undergo functional MR imaging, pre- and post-surgical language evaluation, and electrocortical stimulation mapping. The brain tumor patients will undergo these procedures twice.

SUMMARY:
The purpose of this study is to use an imaging method called functional magnetic resonance imaging (fMRI) in patients who have a tumor near an area of the brain that is believed to control language. The fMRI is a new kind of imaging that uses a strong magnetic field to look at functioning brain tissue. This kind of imaging will be used to study the effect of the brain tumor on your speech.

ELIGIBILITY:
Inclusion Criteria:

* Patient in whom a tumor invades or is directly adjacent to the expected location of one of the language centers.
* At least 18 years of age
* English as first language

Exclusion Criteria:

* Patients with high grade tumors
* History of significant psychiatric condition (e.g. schizophrenia, obsessive-compulsive disorder, significant dementia),
* History of the following neurological conditions: CVA, demyelinating conditions, cerebral palsy, Alzheimer's disease.
* History of significant claustrophobic reactions.
* Pregnancy
* Standard contraindications to MR examinations (e.g. implanted stimulator)
* Patients, who were treated prior to our first scan, will not be eligible to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinics
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2005-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To identify language organization prior to surgery in patients in whom a tumor invades or is directly adjacent to the expected location of one of the language centers. | conclusion of study

SECONDARY OUTCOMES:
To assess language reorganization over time. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Holodny, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org